CLINICAL TRIAL: NCT03907878
Title: A Multi-center, Open-label Study to Investigate the Safety/Tolerability and Efficacy of Ligelizumab (QGE031) in the Treatment of Adult Japanese Patients With Chronic Spontaneous Urticaria (CSU) Inadequately Controlled With H1 Antihistamines
Brief Title: A Safety and Efficacy Study of Ligelizumab in the Treatment of CSU in Japanese Patients Inadequately Controlled With H1- Antihistamines
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CQGE031C1301
Record Dates: First submitted 2019-04-05; First posted 2019-04-09 (Actual); Results first posted 2024-03-08 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Chronic Spontaneous Urticaria
Keywords: CSU; chronic spontaneous urticaria; Japanese; QGE031; Anti-IgE; Ligelizumab; Japan
MeSH Terms: conditions — Chronic Urticaria | interventions — ligelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ligelizumab 120 mg per 1 mL qw4 (Experimental): Subjects received one subcutaneous injection every 4 weeks at 13 visits during the treatment period
  Interventions: Biological: Ligelizumab

INTERVENTIONS:
Biological: Ligelizumab — Liquid in vial
  Other Names: QGE031

SUMMARY:
The purpose of this study was to evaluate the safety and efficacy of ligelizumab in adult Japanese subjects with CSU, who remain symptomatic despite treatment with H1-antihistamines (AHs) at locally approved doses.

The study population consisted of 66 male and female subjects aged ≥ 18 years who were diagnosed with CSU and who remained symptomatic despite the use of H1-AH.

This was a Phase III multi-center, open-label, single arm study. There was a screening period of up to 28 days, a 52 week treatment period, and a 12 week post-treatment follow-up period.

DETAILED DESCRIPTION:
This was a Phase III multi-center, open-label, single arm study. The study consisted of 3 distinct periods:

Screening period (Day -28 to Day -14): Subjects who gave informed consent were assessed for eligibility during this period which lasted for up to 4 weeks.

Treatment period (52 weeks): Subjects had site visits every 4 weeks during this period to receive study drug and complete on-site assessments.

Post-treatment follow-up period (12 weeks): Subject had site visits every 4 weeks with the final visit occurring 16 weeks after the last treatment dose. No study treatment was given during the period.

This study was designed to obtain safety data of QGE031 in 66 Japanese CSU patients.

ELIGIBILITY:
Key Inclusion Criteria:

* Signed informed consent must be obtained prior to participation in the study
* Male and female subjects ≥ 18 years of age at the time of screening
* CSU diagnosis for ≥ 6 months
* Diagnosis of CSU refractory to H1-AH at approved doses at the time of Baseline (Visit 110, Day 1), as defined by all of the following:

  * The presence of itch and hives for ≥ 6 consecutive weeks at any time prior to Visit 1 (Day -28 to Day -14) despite current use of non-sedating H1-AH (at locally approved doses) during this time period
  * UAS7 score (range 0-42) ≥ 16 and HSS7 (range 0-21) ≥ 8 during the 7 days prior to baseline (Visit 110, Day 1)
  * Subjects must be on H1-AH at only approved doses for treatment of CSU for starting at Visit 1 (Day -28 to Day -14)
* Willing and able to complete a daily symptom electronic Diary (eDiary) for the duration of the study and adhere to the study visit schedules

Key Exclusion Criteria:

* History of hypersensitivity to any of the study treatments or excipients or to drugs of similar chemical classes (i.e. to murine, chimeric, or human antibodies)
* Subjects having a clearly defined, predominant trigger of their chronic urticaria (CU) (chronic inducible urticaria (CINDU)) including

  - urticaria factitia (symptomatic dermographism), cold-, heat-, solar-, pressure-, delayed pressure-, aquagenic-, cholinergic-, or contact-urticaria
* Diseases, other than chronic urticaria, with urticarial or angioedema symptoms such as urticarial vasculitis, erythema multiforme, cutaneous mastocytosis (urticaria pigmentosa), and hereditary or acquired angioedema (e.g., due to C1 inhibitor deficiency)
* Subjects with evidence of helminthic parasitic infection as evidenced by stools being positive for a pathogenic organism according to local guidelines. All subjects will be screened at Visit 1. If stool testing is positive for pathogenic organism, the subject will not enter treatment period and will not be allowed to rescreen
* Any other skin disease associated with chronic itching that might influence in the investigator's opinion the study evaluations and results (e.g. atopic dermatitis, bullous pemphigoid (BP), dermatitis herpetiformis, senile pruritus, etc)
* Prior exposure to ligelizumab
* Any H2 antihistamine, Leukotriene Receptor Antagonist (LTRA) (montelukast or zafirlukast) or H1 antihistamines use at greater than approved dose after Visit 1

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2019-04-13 (Actual); Primary Completion 2022-01-26 (Actual); Study Completion 2022-01-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- Japan (10):
  - Novartis Investigative Site, Ichikawa, Chiba
  - Novartis Investigative Site, Obihiro, Hokkaido
  - Novartis Investigative Site, Kobe, Hyōgo
  - Novartis Investigative Site, Nishinomiya, Hyōgo
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Neyagawa, Osaka
  - Novartis Investigative Site, Sakai, Osaka
  - Novartis Investigative Site, Itabashi-ku, Tokyo
  - Novartis Investigative Site, Machida, Tokyo
  - Novartis Investigative Site, Hiroshima

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing access to patient-level data and supporting clinical documents from eligible studies with qualified external researchers. Requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to protect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com
URL: http://www.clinicalstudydatarequest.com

REFERENCES:
- See also: A Plain Language Trial Summary is Available at www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=1387

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 66 participants enrolled at 11 sites in Japan
Pre-assignment Details: Safety Set included all subjects who received at least one dose of study treatment.
Groups:
- Ligelizumab 120 mg Per 1 mL qw4: Subjects received one subcutaneous injection every 4 weeks at 13 visits from baseline to Week 48 during the treatment period. Last treatment was at week 48; and follow up visits were until week 64.
Period: Treatment Period
Arm/Group | Ligelizumab 120 mg Per 1 mL qw4
Started | 66
Completed | 55
Not Completed | 11
Not completed — Withdrawal by Subject | 5
Not completed — Adverse Event | 4
Not completed — Lack of Efficacy | 1
Not completed — Protocol Violation | 1
Period: Follow-up Period
Arm/Group | Ligelizumab 120 mg Per 1 mL qw4
Started | 66
Completed | 60
Not Completed | 6
Not completed — Adverse Event | 3
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Population: Safety Set (SAF) included all subjects who received at least one dose of study treatment.
  Subjects were analyzed according to the study treatment received. Safety Set was used for all safety analyses and also for all efficacy analyses.
Arm/Group | Ligelizumab 120 mg Per 1 mL qw4
Number analyzed (Participants) | 66
Age, Continuous [Mean (Standard Deviation); unit: Years] | 46.4 (13.18)
Age, Customized [Count of Participants; unit: Participants] — Age Categorical
  Participants
    < 18 years | 0
    Between 18 and 65 years | 59
    >=65 years | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53
  Male | 13
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 66

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability of Ligelizumab 120 mg q4w Treatment for 12 Months
Description: Participants with treatment emergent adverse events (AEs) and serious adverse events (SAEs) summary for entire study (64 weeks)
  An AE is any untoward medical occurrence, unfavorable, or unintended sign (including an abnormal laboratory finding), symptom, disease, or injury, temporally associated with the use of a marketed or investigational medicinal product, gene therapy, theragnostic product, or medical device, in patients, clinical-trial subjects, device users, or other persons, whether or not it is considered to be related to or due to the product.
Time Frame: 64 weeks
Population: Safety Set included all subjects who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Ligelizumab 120 mg Per 1 mL qw4
Number analyzed (Participants) | 66
Participants
  Any AEs | 53
  Treatment-related AEs | 11
  Severe AEs | 0
  Moderate AEs | 13
  Deaths | 0
  SAEs | 0
  AEs leading to treatment discontinuation | 4
  SAEs leading to treatment discontinuation | 0

2. Secondary Outcome: UAS7 Change From Baseline Over Time
Description: Mean change from baseline in UAS7 score over time is assessed as absolute change from baseline of UAS7 by visit up to end of study.
  The Urticaria Activity Score (UAS) is the sum of Hive Severity Score (HSS) and Itch Severiry Score (ISS).
  The HSS has a scale of 0 (none) to 3 (> 12 hives/12 hours). A weekly score (HSS7) is derived by adding up the average daily scores of the preceding 7 days. So the range is 0-21; and negative change = improvement.
  The ISS also has a scale of 0 (none) to 3 (severe/difficult to tolerate). A weekly score (ISS7) is derived by adding up the average daily scores of the preceding 7 days. Score range is 0-21; and a negative change from baseline indicates improvement.
  The UAS7 is the sum of the HSS7 score and the ISS7 score, and has a possible range in score of 0-42. A negative change from baseline indicates improvement.
Time Frame: Baseline, Weeks 12, 24, 52, and 64
Population: Safety Set: The number analyzed per row is the number of subjects from the SAF who had a valid assessment for both baseline and the corresponding post baseline time point.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Ligelizumab 120 mg Per 1 mL qw4
Number analyzed (Participants) | 66
Scores on a scale
  Week 12: number analyzed (Participants) | 62
  Week 12 | -18.35 (10.858)
  Week 24: number analyzed (Participants) | 63
  Week 24 | -20.64 (11.082)
  Week 52: number analyzed (Participants) | 56
  Week 52 | -22.92 (11.631)
  Week 64: number analyzed (Participants) | 40
  Week 64 | -15.87 (11.829)

3. Secondary Outcome: HSS7 Change From Baseline Over Time
Description: The HSS has a scale of 0 (none) to 3 (> 12 hives/12 hours):
  0 (None)
  1. (1-6 hives/12 hours)
  2. (7-12 hives/12 hours)
  3. (> 12 hives/12 hours)
  A weekly score (HSS7) is derived by adding up the average daily scores of the preceding 7 days.
  Score range is 0-21; and a negative change indicates improvement.
Time Frame: Baseline, Weeks 12, 24, 52, and 64
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Ligelizumab 120 mg Per 1 mL qw4
Number analyzed (Participants) | 66
Scores on a scale
  Week 12: number analyzed (Participants) | 62
  Week 12 | -10.68 (7.156)
  Week 24: number analyzed (Participants) | 63
  Week 24 | -11.93 (6.815)
  Week 52: number analyzed (Participants) | 56
  Week 52 | -13.33 (6.993)
  Week 64: number analyzed (Participants) | 40
  Week 64 | -9.29 (7.136)

4. Secondary Outcome: ISS7 Change From Baseline Over Time
Description: The ISS has a scale of 0 (none) to 3 (severe):
  0 None
  1. Mild (minimal awareness, easily tolerated)
  2. Moderate (definite awareness, bothersome but tolerable)
  3. Severe (difficult to tolerate)
  The ISS also has a scale of 0 (none) to 3 (severe/difficult to tolerate). A weekly score (ISS7) is derived by adding up the average daily scores of the preceding 7 days. So the score range of ISS7 is 0-21; and a negative change from baseline indicates improvement.
Time Frame: Baseline, Weeks 12, 24, 52, and 64
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Ligelizumab 120 mg Per 1 mL qw4
Number analyzed (Participants) | 66
Scores on a scale
  Week 12: number analyzed (Participants) | 62
  Week 12 | -7.68 (4.376)
  Week 24: number analyzed (Participants) | 63
  Week 24 | -8.72 (5.054)
  Week 52: number analyzed (Participants) | 56
  Week 52 | -9.59 (5.434)
  Week 64: number analyzed (Participants) | 40
  Week 64 | -6.58 (5.473)

5. Secondary Outcome: Percentage of Participants Who Achieved the Complete UAS7 = 0 Response Over Time
Description: Assessed as the proportion of subjects achieving UAS7 = 0 over time.
  The UAS7 has a possible range in score of 0-42, and its complete response (complete urticaria control) was defined as UAS7 = 0
Time Frame: Weeks 12, 24, 52, and 64
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Ligelizumab 120 mg Per 1 mL qw4
Number analyzed (Participants) | 66
Participants
  Week 12: number analyzed (Participants) | 62
  Week 12 | 14
  Week 24: number analyzed (Participants) | 63
  Week 24 | 26
  Week 52: number analyzed (Participants) | 56
  Week 52 | 28
  Week 64: number analyzed (Participants) | 40
  Week 64 | 11

6. Secondary Outcome: Percentage of Participants Who Achieved the Complete HSS7 = 0 Response Over Time
Description: The proportion of subjects achieving HSS7 = 0 (complete absence of hives) over time
  The HSS has a scale of 0 (none) to 3 (> 12 hives/12 hours). A weekly score (HSS7) is derived by adding up the average daily scores of the preceding 7 days. So the range is 0-21; and negative change = improvement.
Time Frame: Weeks 12, 24, 52, and 64
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Ligelizumab 120 mg Per 1 mL qw4
Number analyzed (Participants) | 66
Participants
  Week 12: number analyzed (Participants) | 62
  Week 12 | 17
  Week 24: number analyzed (Participants) | 63
  Week 24 | 31
  Week 52: number analyzed (Participants) | 56
  Week 52 | 33
  Week 64: number analyzed (Participants) | 40
  Week 64 | 13

7. Secondary Outcome: Percentage of Participants Who Achieved the Complete ISS7 = 0 Response Over Time
Description: The ISS also has a scale of 0 (none) to 3 (severe/difficult to tolerate). A weekly score (ISS7) is derived by adding up the average daily scores of the preceding 7 days. Score range is 0-21; and a negative change from baseline indicates improvement.
Time Frame: Weeks 12, 24, 52, and 64
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Ligelizumab 120 mg Per 1 mL qw4
Number analyzed (Participants) | 66
Participants
  Week 12: number analyzed (Participants) | 62
  Week 12 | 14
  Week 24: number analyzed (Participants) | 63
  Week 24 | 27
  Week 52: number analyzed (Participants) | 56
  Week 52 | 30
  Week 64: number analyzed (Participants) | 40
  Week 64 | 12

8. Secondary Outcome: Change From Baseline in the Dermatology Life Quality Index (DLQI)
Description: Assessed by absolute change from baseline of DLQI up to end of study. Score range is from 0-30:
  0-1 No effect on patients life 2-5 Small effect on patients life 6-10 Moderate effect on patients life 11-20 Very large effect on patients life 21-30 Extremely large effect on patients life
  A negative change indicates improvement.
Time Frame: Baseline, Weeks 12, 24, 52 and 64
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Ligelizumab 120 mg Per 1 mL qw4
Number analyzed (Participants) | 66
Scores on a scale
  Week 12: number analyzed (Participants) | 64
  Week 12 | -6.66 (4.870)
  Week 24: number analyzed (Participants) | 61
  Week 24 | -6.39 (6.127)
  Week 52: number analyzed (Participants) | 64
  Week 52 | -6.69 (5.858)
  Week 64: number analyzed (Participants) | 59
  Week 64 | -5.78 (5.474)

9. Secondary Outcome: Percentage of Participants Who Achieved Dermatology Life Quality Index (DLQI) = 0/1 by Visit up to End of Study
Description: Percentage of participants who achieved DLQI = 0/1 by visit up to end of study, assessed by absolute change from baseline of DLQI up to end of study. Score range is from 0-30:
  0-1 No effect on patients life 2-5 Small effect on patients life 6-10 Moderate effect on patients life 11-20 Very large effect on patients life 21-30 Extremely large effect on patients life
  A negative change indicates improvement.
Time Frame: Weeks 12, 24, 52, and 64
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Ligelizumab 120 mg Per 1 mL qw4
Number analyzed (Participants) | 66
Participants
  Week 12: number analyzed (Participants) | 64
  Week 12 | 37
  Week 24: number analyzed (Participants) | 61
  Week 24 | 40
  Week 52: number analyzed (Participants) | 64
  Week 52 | 44
  Week 64: number analyzed (Participants) | 59
  Week 64 | 30

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) and Serious Adverse Events were collected after signature of the informed consent form until the end of study at 64 weeks.
Description: An AE is any untoward medical occurrence, unfavorable, or unintended sign (including an abnormal laboratory finding), symptom, disease, or injury, temporally associated with the use of a marketed or investigational medicinal product, gene therapy, theragnostic product, or medical device, in patients, clinical-trial subjects, device users, or other persons, whether or not it is considered to be related to or due to the product.
Groups:
- QGE031 120mg: Ligelizumab 120 mg per 1 mL qw4
Arm/Group | QGE031 120mg
All-Cause Mortality (participants affected / at risk) | 0/66
Serious Adverse Events (participants affected / at risk) | 0/66
Other Adverse Events (participants affected / at risk) | 41/66
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | QGE031 120mg (N=66)
Abdominal pain upper (Gastrointestinal disorders) | 2
Dental caries (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 2
Injection site erythema (General disorders) | 3
Injection site pain (General disorders) | 2
Injection site reaction (General disorders) | 2
Malaise (General disorders) | 2
Pyrexia (General disorders) | 6
Hepatic function abnormal (Hepatobiliary disorders) | 2
Cystitis (Infections and infestations) | 3
Folliculitis (Infections and infestations) | 2
Gastroenteritis (Infections and infestations) | 2
Influenza (Infections and infestations) | 3
Nasopharyngitis (Infections and infestations) | 8
Oral herpes (Infections and infestations) | 2
Arthropod bite (Injury, poisoning and procedural complications) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 5
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Carpal tunnel syndrome (Nervous system disorders) | 2
Headache (Nervous system disorders) | 4
Hypoaesthesia (Nervous system disorders) | 2
Acne (Skin and subcutaneous tissue disorders) | 3
Asteatosis (Skin and subcutaneous tissue disorders) | 2
Dermatitis contact (Skin and subcutaneous tissue disorders) | 5
Eczema (Skin and subcutaneous tissue disorders) | 9
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 2
Urticaria (Skin and subcutaneous tissue disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2020-02-14): https://cdn.clinicaltrials.gov/large-docs/78/NCT03907878/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-22): https://cdn.clinicaltrials.gov/large-docs/78/NCT03907878/SAP_001.pdf